CLINICAL TRIAL: NCT05388292
Title: Effect of Computer-based Decision Support System on Emergency Triage Management
Brief Title: Decision Support System on Emergency Triage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Songül BİŞKİN ÇETİN, Principal Investigator, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2012-KAEK-20-2019
Record Dates: First submitted 2022-04-28; First posted 2022-05-24 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Triage; Emergencies; Decision Support Systems
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Masking Description: This is a quasi-experimental study with a single-group pre-test and post-test design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Development of triage decision support system (Other): This is a quasi-experimental study with a single-group pre-test and post-test design.
  The study consisted of three stages. In the first stage, a structured Query Language Script was developed to evaluate the accuracy and duration of pre-and post-DSS triage decisions. In the second stage (pre-test), the accuracy and duration of pre-DSS triage decisions were evaluated. In the second stage, a DSS was prepared with rule-based decision trees method using the ESI and ATS algorithms and was integrated into the HIMS. In the third and last stage (post-test), the effect of the developed Emergency Triage Decision Support System on triage management was evaluated against the accuracy and duration of triage decisions.
  Interventions: Other: Emergency triage decision support system

INTERVENTIONS:
Other: Emergency triage decision support system — Evaluating the impact of the developed Emergency Triage Decision Support System on triage management

SUMMARY:
The objective of this study is to design a computer-based Decision Support System (DSS) using the ESI (Emergency Severity Index) and ATS (Australasian Triage Scale) algorithms, integrate it into the Hospital Information Management System (HIMS), evaluate the effect of the triage management in the emergency department and ensure the continuity of the system.

DETAILED DESCRIPTION:
Background: Triage in the emergency department overstrains employees due to patient density, diversity, and time pressure.

Aim: The objective of this study is to design a computer-based Decision Support System (DSS) using the ESI (Emergency Severity Index) and ATS (Australasian Triage Scale) algorithms, integrate it into the Hospital Information Management System (HIMS), evaluate the effect of the triage management in the emergency department and ensure the continuity of the system.

Study design: This is a quasi-experimental study with a single-group pre-test and post-test design. The study consisted of three stages.

Methods: In the first stage, a SQL (Structured Query Language) Script was developed to evaluate the accuracy and duration of pre-and post-DSS triage decisions. In the second stage (pre-test), the accuracy and duration of pre-DSS triage decisions were evaluated. In the second stage, a DSS was prepared with rule-based decision trees method using the ESI and ATS algorithms and was integrated into the HIMS. In the third and last stage (post-test), the effect of the developed Emergency Triage Decision Support System (ETDSS) on triage management was evaluated against the accuracy and duration of triage decisions.

ELIGIBILITY:
Inclusion Criteria:

Data of adult patients who applied to the adult emergency department and whose triage record was opened by a triage nurse.

Patient data with no probable or definitive diagnosis of COVID-19.

Exclusion Criteria:

Data of pediatric trauma patients (under 18 years of age) Patient data for which the triage record was opened by non-nursing healthcare professionals Patient data recorded in triage by nurses who did not receive ATKDS, Emergency nurse triage, ESI, ATS training Data of patients who applied with a probable/definite diagnosis of COVID-19 and underwent PCR testing Patient data in the date range when extraordinary changes were made in the adult emergency department patient triage area and evaluation process due to the COVID 19 pandemic and the developed system could not be used (must use the SB COVID Algorithm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5038 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Emergency Triage Decision Support System triage management was evaluated against the accuracy and duration of triage decisions | 8 weeks (triage decision' accuracy in eight-week hospital information management system data)
  The effect of the decision support system on the triage decision accuracy

SECONDARY OUTCOMES:
Emergency Triage Decision Support System | 8 weeks (triage decision' duration in eight-week hospital information management system data)
  The effect of decision support system on triage decision duration

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Cebeci, Study Chair — 1962
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No